CLINICAL TRIAL: NCT00744250
Title: Intraduodenal Aspiration Study to Assess the Bioavailability of Oral Pancrecarb® Compared to Placebo Control in Patients With Pancreatic Insufficiency
Brief Title: Intraduodenal Aspiration Study to Assess the Bioavailability of Oral Pancrecarb® Compared to Placebo Control
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No longer required study by FDA for NDA approval.
Sponsor: Digestive Care, Inc. (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCRC-2712; 08-0819
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Exocrine Pancreatic Insufficiency; Chronic Pancreatitis; Cystic Fibrosis
Keywords: Exocrine Pancreatic Insufficiency; Chronic Pancreatitis; Cystic fibrosis; Pancrelipase; Pancrecarb; Intraduodenal aspiration; Bioavailability
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic; Cystic Fibrosis | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Pre-treatment vs. post-treatment-
  In the first phase, before administration of the capsules and liquid diet, baseline gastric and duodenal secretions will be aspirated via the oro-enteric tube. Subjects will get 5 placebo capsules at Time=0 given orally with the liquid Lundh diet. Pancreato-biliary and duodenal secretions in the duodenal region will be aspirated continuously over the first 20 min. Gastric and duodenal fluids will be aspirated from 20-180 min at specified time points. Following a rest of 1 hour, the same process will be repeated with the drug capsules. At the end of the study the catheter will be removed and patient will be offered a meal.
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase — PANCRECARB MS-16
  Other Names: Pancrecarb®

SUMMARY:
The purpose of this research study is to learn about the activity of oral Pancrecarb® (a pancreatic enzyme preparation which contains proteins that help to digest food), administered by mouth as a capsule filled with specially coated granules in patients taking exogenous pancreatic enzyme therapy. Specific enzymes activities will be determined from samples of stomach and intestinal fluids after a standard liquid meal.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to assess the bioavailability of oral Pancrecarb® (exogenous pancreatic enzyme administered orally as a capsule filled with enteric coated granules) compared to placebo control in patients with pancreatic insufficiency. Lipase, amylase and protease activities will be determined from stomach and duodenal aspirates after standard meal stimulation.

Participants:

Patients with pancreatic insufficiency will be recruited as the study population.

Procedures (methods):

Eligible subjects will undergo an initial screening phase and will provide a stool sample to confirm pancreatic exocrine insufficiency based on a spot fecal elastase-1 of < 75 mcg/g stool. Within one month after the screening phase, subjects meeting inclusion criteria will be scheduled to arrive in the GCRC by 7pm. If the subject is a female of child bearing age, a serum pregnancy test will be checked. At 7am the subject will be escorted to fluoroscopy for placement of an oro-enteric tube. Once the tip of the tube has been positioned in the duodenum, the subject will be escorted back to the GCRC. Prior to administration of the capsules and liquid diet, baseline gastric and duodenal secretions will be aspirated via the oro-enteric tube by the investigators. Subjects will then receive 5 capsules of active drug with a standard liquid Lundh diet of 360 mL over a 10 minute period, administered to simulate a fed state. Then duodenal and gastric secretions will be aspirated from the tube over a 3-hour period. At the end of the 3 hours, the subject will be allowed to rest for 60 minutes. The second phase will consist of 5 capsules of placebo again with a standard liquid Lundh diet , and another 3-hour aspiration phase. After the second 3-hour aspiration period, the balloon will be deflated and the tube will be removed. Subjects will be observed for 30 minutes and then discharged.

ELIGIBILITY:
Inclusion Criteria:

* Documented pancreatic enzyme insufficiency as determined by spot fecal elastase-1 (<75 mcg/g) at the time of screening
* Required daily exogenous enzyme supplementation with commercially available pancreatic enzymes
* ≥ 18 years of age
* Male and female subjects
* Able to swallow capsules
* Clinically stable with no evidence of an acute medical conditions

Exclusion Criteria:

* History of fibrosing colonopathy in cystic fibrosis subjects
* Current diagnosis or a history of distal intestinal obstruction syndrome (DIOS) in the past 4 months
* Known contraindications, sensitivity or hypersensitivity to porcine pancreatic enzymes, benzocaine or similar products
* Women with a positive serum beta-hCG at the time of screening or the day of the study (due to radiation exposure)
* Liver disease
* ALT or AST ≥ 3 time the upper limit of normal
* Bilirubin ≥ 3 times the upper limit of normal
* Acute pancreatitis or acute exacerbation of chronic pancreatitis within 90 days
* Use of medications which affect with intestinal transit (example, narcotics, erythromycin, metoclopramide etc.)
* Subjects receiving treatment with antacids, H2 receptor blockers, or proton pump inhibitors and unable to discontinue these within 72 hr prior to the study day
* Diabetes mellitus
* A medical condition which the investigator deems significant enough to interfere with the ability of the subject to participate in the intubation study or interfere with the assessment of enzyme bioavailability
* Small bowel disease (i.e. celiac disease)
* Lactose intolerance
* History of gastric resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Peak levels of three enzymes - lipase, amylase, and protease - each measured in U/ml will be outcomes | Samples will be collected over two consecutive 3 hour study periods and sent for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gangarosa, M.D., Principal Investigator — University of North Carolina, Chapel Hill; Kim Brouwer, PharmD, PhD, Principal Investigator — UNC School of Pharmacy
Locations (1):
- UNC Healthcare, Chapel Hill, North Carolina, United States